CLINICAL TRIAL: NCT05503667
Title: Neoadjuvant Furmonertinib Plus Bevacizumab or Furmonertinib Monotherapy for Resectable and Potentially Resectable Stage III-IVA EGFR Mutation-Positive Lung Adenocarcinoma: A Randomized, Controlled, Open-label, Single-center Phase II Clinical Trial
Brief Title: Neoadjuvant Furmonertinib Plus Bevacizumab or Furmonertinib Monotherapy for Resectable and Potentially Resectable Stage III-IVA EGFR Mutation-Positive Lung Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Peng Zhang, Director of science and education department, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LungMate-012
Record Dates: First submitted 2022-08-13; First posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Lung Adenocarcinoma Stage III; Lung Adenocarcinoma Stage IV; EGFR Gene Mutation
Keywords: neoadjuvant chemoimmunotherapy
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — aflutinib; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Furmonertinib Plus Bevacizumab (Experimental): Furmonertinib Plus Bevacizumab
  Interventions: Drug: Furmonertinib; Drug: Bevacizumab
- Furmonertinib (Active Comparator): Furmonertinib monotherapy
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — Furmonertinib 80 mg/day for 16 weeks
  Other Names: Ivesa
Drug: Bevacizumab — bevacizumab 400 mg/4 weeks i.v. for 4 times
  Other Names: Avastin
  Arms: Furmonertinib Plus Bevacizumab

SUMMARY:
To explore the efficacy and safety of neoadjuvant furmonertinib combined with bevacizumab in the treatment of resectable and potentially resectable stage III-IVA EGFR mutation-positive lung adenocarcinoma.

DETAILED DESCRIPTION:
The best treatment for lung cancer is still radical resection, which is indicated for stage I-II and some stage III patients, but surgery is only suitable for 20-25% of NSCLC patients. Furmonertinib is a third-generation TKI drug. Compared with first and second-generation TKI drugs, it has good benefits in the Chinese population, patients with brain metastases, and patients with 19del/L858R mutation, with better and longer-lasting effects, and can significantly improve the progression-free survival of patients. Neoadjuvant therapy can shrink the tumor, increase the rate of complete surgical resection, remove micrometastases, and reduce the risk of recurrence. Cases of patients with locally advanced (IIIA-N2) NSCLC have been reported with neoadjuvant TKI therapy, and it has been found that neoadjuvant TKI therapy can downgrade or even complete tumor remission. However, for locally advanced potentially resectable, or EGFR mutation-positive NSCLC patients with single-organ metastasis, the efficacy of third-generation EGFR-TKI combined with VEFGR inhibitor combined with targeted therapy after induction and surgery is still unclear. Limited clinical research data suggest that this new treatment mode (induction therapy-surgery-adjuvant therapy) can significantly improve the progression-free survival of patients. However, the overall survival rate under the new treatment mode and the promotion of clinical work urgently need higher-level clinical evidence to support clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Lung adenocarcinoma patient with EGFR sensitive mutation as confirmed by needle biopsy;
* At stage III-IVA (TNM Staging, Version 8) as identified by chest CT, PET-CT or/and EBUS;
* No systemic metastasis (confirmed by head MRI, whole body bone scan, PET-CT, liver and adrenal CT, etc.);
* With the feasiblility or potential feasibility to receive radical surgery (radical lung lobectomy+systematic lymph node dissection);
* Good lung function that could tolerate surgical treatment;
* Aged >= 18 years;
* At least one measurable tumor foci (the longest diameter measured by CT shall be > 10 mm);
* Other major organs shall function well (liver, kidney, blood system, etc.):
* ECOG PS score shall be 0-1;
* The child-bearing female must undergo pregnancy test within 7 days before starting the treatment and the result shall be negative. Reliable contraceptive measures, such as intrauterine device, contraceptive pill and condom, shall be adopted during the trial and within 30 days after completion of the trial. The child-bearing male shall use condom for contraception during the trial and within 30 days after completion of the trial;
* The patient shall sign the Informed Consent Form.

Exclusion Criteria:

* The patient has undergone any systemic anti-cancer treatment for NSCLC, including cytotoxic drug treatment, targeted drug treatment and experimental treatment, etc.;
* The patient suffers from any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina pectoris, angina pectoris that starts to attack within the last 3 months, congestive heart failure [≥ Grade II specified by New York Heart Association (NYHA)], cardiac infarction (6 months before enrollment), severe arrhythmia and liver, kidney or metabolic diseases that requires drug treatment;
* The patient is a carrier of HIV;
* The patient is currently suffering from interstitial lung disease;
* The patient had undergone other major systemic operations or suffered from severe trauma within 3 months before the trial;
* The patient is allergic to furmonertinib or its any excipients;
* The patient is allergic to bevacizumab or its any excipients;
* The female patient is in pregnancy or lactation period;
* There are any conditions under which the investigator considers the patient is not suitable to be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 21 months
  It refers to the proportion of patients who have had a complete response or partial response (according to RECIST1.1) as confirmed by CT evaluation after 3 weeks in all patients who have completed the neoadjuvant therapy. Only patients with measurable lesions at baseline will be analyzed.

SECONDARY OUTCOMES:
Disease-free survival (DFS) | up to 54 months
  It refers to the time from radical surgery to relapse or death of a participant due to disease progression. In the case of a patient who still survives at the time of analysis, the latest evaluation date will be used for interpolation (censoring).
Overall survival (OS) | up to 60 months
  It is defined as the time from enrollment to death of participant due to any cause. In the case of a patient who still survives at the time of analysis, the date of last contact will be taken as the censoring date. In the event of a patient with the survival status unknown, the date when the patient is last known to be alive will be used for interpolation (censoring).
Health related quality of life (HRQol) | up to 6 months
  The assessment is made according to the Quality of Life Scale for Lung Cancer Patients (EORTC-QLQ-C30 & LC13, Version 3). EORTC's QLQ-C30 & LC13 (V3.0) is a core scale for lung cancer patients, with a total of 43 items. Among them, Item 29 and 30 are divided into seven grades, which are assigned with 1 to 7 scores according to the answer options. The other items are divided into 4 grades: Not at All, A Little, Quite a Bit, and Very Much, assigned with 1 to 4 scores respectively. The higher score, the worse quality.
Progression-free survival (PFS) | up to 54 months
  It refers to the time from the first administration of SHR1316 in this study to the disease progression or death (including any cause of death in the case of no progression) , regardless of whether the patient exits from the treatment or receives other anti-cancer treatment before progression.
R0 resection | up to 24 months
  It is defined as the proportion of patients with negative surgical margin and no residual found under microscope after resection in all patients who have completed the treatment.
Pathological downstaging rate | up to 24 months
  It is defined as the proportion of patients who have completed the 8-week treatment with afatinib before operation and have achieved a T stage downing of the tumor as confirmed by CT evaluation after 3 weeks in all patients who have completed the treatment.
Treatment-related adverse events (AEs) | up to 6 months
  It refers to the number of adverse events related to furmonertinib plus bevacizumab therapy or furmonertinib monotherapy as evaluated according to CTCAE v4.0.
Pathological complete response rate (pCR) | up to 24 months
  It refers to the number of cases with no residual invasive cancer in the primary tumor and lymph node HE staining accounted for the proportion of all patients who completed the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No